CLINICAL TRIAL: NCT04069442
Title: cDC1 Prognostic and Predictive Role in Non-Small-Cell Lung Cancer Patients Receiving Immune Checkpoint Inhibitors
Acronym: LUNG-PREDICT
Status: Withdrawn | Type: Observational
Why Stopped: access to human body samples by another existing cohort
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.100; 2019-A00959-48 (Other: ID RCB)
Record Dates: First submitted 2019-08-12; First posted 2019-08-28 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cDC-1 positive: cDC-1 positive patients according to RNAseq and in situ analysis
  Interventions: Other: This is a non-interventional study
- cDC-1 negative: cDC-1 negative patients according to RNAseq and in situ analysis
  Interventions: Other: This is a non-interventional study

INTERVENTIONS:
Other: This is a non-interventional study — This is a non-interventional study

SUMMARY:
The response rate of immune checkpoint inhibitors remains relatively low and the identification of the new predictive biomarkers is necessary. The rare population of cDC1 is very interesting, as its mouse counterparts is essential for the cross presentation of tumor-associated antigens, tumor immunity and response to immunotherapies. Their role in humans has not been studied. This proposal aims to study the prognostic role of cDC1 in a cohort of patients with advanced NSCLC, possibly demonstrating their positive predictive value of immune checkpoint inhibitors response.

DETAILED DESCRIPTION:
Multicenter study aiming to collect patient's clinical data retrospectively and their histological samples prospectively.

The cohort will include:

* 30 patients PD-L1 > 50% treated with pembrolizumab in first line and having a progression free survival ≥ 3 months
* 30 patients PD-L1 > 50% treated with pembrolizumab in first line and having a progression free survival < 3 months
* 30 patients PD-L1 < 50% treated with cisplatin-based chemotherapy in first line

ELIGIBILITY:
Inclusion Criteria:

* NSCLC diagnosis
* Advanced disease (Stage III-IV) according to the TNM 7th/8th classification
* Patients have to have performed pembrolizumab in first line if PD-L1 ≥ 50% or cisplastin-based chemotherapy if PD-L1 < 50%
* FFPE material available from diagnostic sample

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort of pembrolizumab or cisplatin-based chemiotherapy treated patients performing these regimens in first-line according to their PD-L1 score
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 1 year
  To validate the cDC1 infiltration as predictive biomarker of pembrolizumab response

SECONDARY OUTCOMES:
Overall response rate (ORR) | 1 year
  To compare the overall response rate (ORR) of cDC1-positive patients to cDC1 negative ones within those treated with pembrolizumab and on the entire cohort
Time to treatment failure (TTF) | 1 year
  To compare the time of treatment failure (TTF) on CDC1-positive patients to negatives ones within those treated with pembrolizumaband on the entire cohort

OTHER OUTCOMES:
Overall survival (OS) | 1 year
  To compare the overall survival (OS) of cDC1-positives patients to negatives ones within those treated with pembrolozumab and on the entire cohort

CONTACTS AND LOCATIONS:
Overall Officials: Elisa GOBBINI, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble-Alpes, Grenoble, Isère, France